CLINICAL TRIAL: NCT02780544
Title: Is There a Difference in Pain Score, Stress Response and Motor Repertoire in Infants Given Skin-to-skin Contact With the Mother/Father or Standard Care During Screening for Retinopathy?
Brief Title: Infant-parent Skin-to-skin Contact During Screening for Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011/2532b
Record Dates: First submitted 2016-05-12; First posted 2016-05-23 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Retinopathy of Prematurity
Keywords: Infant, premature; Pain; Stress, physiological; Stress, psychological; skin-to-skin contact
MeSH Terms: conditions — Retinopathy of Prematurity; Premature Birth; Pain; Stress, Psychological | interventions — Incubators; Sucrose

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- skin-to-skin contact + sucrose (Experimental): the infants get 2 eye examinations within 1 week in randomized order, one in skin-to-skin position with a parent (intervention group) and one in the incubator (standard care). Sucrose (0.2 ml) lingual will be given for pain relief according to standard care two minutes before either eye examination.
  Interventions: Behavioral: skin-to-skin contact; Drug: Sucrose
- incubator + sucrose (Active Comparator): the infants get 2 eye examinations within 1 week in randomized order, one in the incubator (standard care) and one in skin-to-skin position with a parent (intervention group). Sucrose (0.2 ml) lingual will be given for pain relief according to standard care two minutes before either eye examination
  Interventions: Device: incubator; Drug: Sucrose

INTERVENTIONS:
Behavioral: skin-to-skin contact — skin-to-skin contact with parent during eye examination.
  Arms: skin-to-skin contact + sucrose
Device: incubator — staying in incubator during eye examination.
  Arms: incubator + sucrose
Drug: Sucrose — oral sucrose before eye examination

SUMMARY:
Retinopathy of prematurity (ROP) is a feared complication of premature birth. If discovered in time, the disease can be treated, and impaired vision or blindness can be reduced. Premature infants are therefore examined regularly after birth. However, the examination is painful and stressful for the infant. Painful experiences might lead to a pathological stress response later in life and should therefore be prevented.

In this study skin-to-skin contact with a parent is tested for relief of pain and stress in preterm infants being examined for retinopathy of prematurity.

ELIGIBILITY:
Inclusion Criteria:

* Infants < 32 weeks of gestational age (< 31+6 weeks)

Exclusion Criteria:

* Infants with ongoing analgesic treatment

Ages: 31 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
pain score | during eye examination
  Premature Infant Pain Profile (PIPP): score range 0-21. Assessed during and immediately after completed examination). PIPP scoring via video recording by an external observer (blinded)

SECONDARY OUTCOMES:
cortisol in saliva | 60 minutes after eye examination
  to measure stress response
General movements | in 5 minutes after eye examination
  Prechtl method on the General Movements Assessment (GMA) and classified according to the general movements optimality list for preterm general movements and writing movements

CONTACTS AND LOCATIONS:
Overall Officials: Hakon Bergseng, PhD, Principal Investigator — St. Olavs University Hospital
Locations (1):
- St.Olavs University Hospital, Trondheim, Trøndelag, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kristoffersen L, Stoen R, Bergseng H, Follestad T, Theodorsson E, Vederhus B, Adde L, Austeng D. Skin-to-skin contact during eye examination did not reduce pain compared to standard care with parental support in preterm infants. Acta Paediatr. 2019 Aug;108(8):1434-1440. doi: 10.1111/apa.14699. Epub 2019 Jan 18. PMID 30561825